CLINICAL TRIAL: NCT00079586
Title: A Study Comparing Angiomax (Bivalirudin) to Heparin With Protamine Reversal in Patients Undergoing Cardiac Surgery on Cardiopulmonary Bypass (CPB)
Brief Title: Comparing Angiomax to Heparin With Protamine in Patients Undergoing Cardiopulmonary Bypass (CPB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-06; EVOLUTION-On
Record Dates: First submitted 2004-03-09; First posted 2004-03-11 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Heparin; bivalirudin

ARMS (2):
- Heparin (Active Comparator): unfractionated heparin will be administered as per institutional practice
  Interventions: Drug: Heparin
- Angiomax (Experimental): 1.0 mg/kg IV bolus followed by a 2.5 mg/kg/hr IV infusion
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Heparin — Unfractionated Heparin per institutional practice
  Arms: Heparin
Drug: Bivalirudin — 1.0 mg/kg IV bolus followed by a 2.5 mg/kg/hr IV infusion
  Arms: Angiomax

SUMMARY:
The purpose of this study is to demonstrate that in patients undergoing coronary artery bypass grafting (CABG) or CABG-Valve, or Isolated Cardiac Valve surgery on CPB (cardiac surgery), Angiomax is a safe and effective alternative anticoagulant to heparin with protamine reversal.

ELIGIBILITY:
Inclusion Criteria

* Provide written informed consent before initiation of any study related procedures.
* Be at least 18 years of age.
* Be scheduled for CABG, CABG and single valve surgery, or isolated single valve surgery on CPB. Patients undergoing repeat (redo) CABG are also considered eligible for this study.

Exclusion Criteria

* Confirmed pregnancy at time of randomization via IVRS (if woman of child-bearing potential) (Urine or serum pregnancy test)
* Cerebrovascular accident within 6 months, or any cerebrovascular accident with a residual neurological deficit.
* Intracranial neoplasm, arteriovenous malformation or aneurysm.
* Dependency on renal dialysis or creatinine clearance <30 mL/min.
* Ongoing treatment with warfarin (or other oral anticoagulant) at the time of randomization.

Patients previously treated with warfarin may be enrolled if warfarin therapy can be safely discontinued and baseline INR is < 1.3 times control in the absence of heparin therapy.

* Known allergy to Angiomax or hirudin-derived drugs, or known sensitivity to any component of the product.
* Patients receiving clopidogrel (Plavix®) within the previous 5 days of randomization
* Patients receiving a glycoprotein IIb/IIIa inhibitor within the previous 48 hours if abciximab (ReoPro®) or 24 hours if eptifibatide (Integrilin®) or tirofiban (Aggrastat®) of randomization.
* Patients receiving lepirudin (Refludan®) or argatroban within the previous 24 hours prior to randomization.
* Patients receiving LMWH or thrombolytics within the previous 12 hours or unfractionated heparin within 30 minutes of randomization.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of randomization.
* Refusal to undergo blood transfusion should it become necessary.
* Any other disease or condition, which, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the trial.
* Planned surgical procedure in which proximal anastomoses will precede distal anastomoses of the bypass grafts.
* Planned (>1) double (or greater) valve repair-replacement (e.g.: AVR-MVR) surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04; Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Lloyd, MD, Study Director — The Medicines Company
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States